CLINICAL TRIAL: NCT07186946
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Comparative Bioavailability (Unblinded) of THRV-1268 in Health Obese Adult Participants
Brief Title: Phase 1, Single Ascending Dose Study to Evaluate the Safety, Tolerability, PK, PD, and Comparative Bioavailability of THRV-1268 in Obese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thryv Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: THRV-1268-0369
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: heart failure; obesity; cardiometabolic; atrial fibrillation
MeSH Terms: conditions — Heart Failure; Obesity; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In period 2 of cohort 1, relative bioavailability is unmasked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) THRV-1268 low dose (100mg) (Experimental): In Period 1 of cohort 1 will receive a single oral dose of THRV-1268 100mg
  Interventions: Drug: THRV-1268; Drug: Placebo
- THRVY-1268 high dose (200mg) (Experimental): In cohort 2, will receive a single oral dose of THRV-1268 200mg
  Interventions: Drug: THRV-1268; Drug: Placebo

INTERVENTIONS:
Drug: THRV-1268 — THRV-1268 a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
Drug: Placebo — Placebo

SUMMARY:
A research study that involves the use of an investigational drug called THRV-1268. The main purpose is to measure the safety (whether it causes any side effects) and tolerability (if it does cause any side effects, how well your body is able to handle them) in healthy obese adults. This study will also look at how the drug moves through the body, is absorbed, distributed, metabolized and eliminated.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated Informed Consent Document (ICD).
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Healthy adult male or female participants.
* If female, meets one of the following criteria:

  1. Women of childbearing potential (WOCBP) who agrees to use any of the acceptable contraceptive methods:

     1. Abstinence from heterosexual intercourse from Screening through at least 30 days from last study dose.
     2. One of the following highly-effective contraception methods:

        1. intrauterine device (with or without hormones) used from at least 28 days prior to Screening through to at least 30 days from last study dose
        2. male partner vasectomized at least 6 months prior to Screening visit
     3. Double-barrier contraception method (e.g., condom and spermicide) used from 28 days prior to Screening through at least 30 days from last study dose Or
  2. Physiological postmenopausal status, defined as the absence of menses for at least 12 months following cessation of all exogenous hormonal treatments (without an alternative medical condition) at Screening and prior to the first study drug administration.

     Or
  3. Surgically sterile, defined as those who have had hysterectomy, bilateral oophorectomy and/or bilateral salpingectomy, or bilateral tubal ligation/occlusion.
* Male volunteers agree to use a double-barrier method (e.g., condom and spermicide) or agree to remain abstinent from heterosexual intercourse at the time of Screening, during the study, and for 90 days following the study dose. Men who are biologically capable of fathering children must also agree to refrain from sperm donation for the duration of the treatment period and for at least 90 days after the last study dose.
* Aged at least 18 years but not older than 55 years (both years inclusive) at screening.
* Body mass index (BMI) more than or equal to 30.0 kg/m2 and up to 40.0 kg/m2 (both inclusive).
* Body weight ≥ 90.0 kg.
* Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 90 days prior to the first study drug administration).
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings in the physical examination (including vital signs), safety clinical laboratory tests, and/or ECG, as determined by an Investigator.
* Ability to swallow whole tablets.

Exclusion and Restriction Criteria

* Clinically significant cardiovascular, gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, or psychiatric disease, or any other condition, which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study results.
* Female who is lactating.
* Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration or planning to be pregnant.
* Male participants with a history of oligospermia or azoospermia or any other disorder of the reproductive system.
* Male participants who are undergoing treatment or evaluation for infertility.
* The average of 3 BP measurements performed after resting supine quietly for at least 5 min, and approximately 1 min between each measurement:
* Screening or baseline (Day -1, Period 1) :

  1. systolic BP <100 mmHg or >145 mmHg;
  2. diastolic BP <50 mmHg or >95; or
  3. pulse rate ≤ 50 beats per minute (bpm) using a validated digital BP device.
* These can be repeated in triplicate once after an additional quiet resting period.
* Orthostatic BP performed after at least 5 mins in supine position and then after standing for at least 2 minutes but no more than 3 minutes with a reduction in systolic BP >20 mmHg, or a reduction in diastolic BP >10 mmHg, using a validated digital BP device.
* History of significant hypersensitivity to THRV-1268, kinase inhibitors or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Screening and check-in at Period 1: 12-lead ECG demonstrating at least one of the following:

  1. Heart rate ≤50 bpm or >100 bpm.
  2. PR interval >200 ms;
  3. QRS duration >110 ms, or
  4. QTcF ≥ 450 ms in males and 470 ms in females;
  5. atrioventricular block; branch bundle block, significant ST T wave abnormalities or flat T waves that could interfere with QT analysis
* History or evidence of any of the following: myocardial infarction; cardiac valvulopathy; cardiac surgery revascularization (coronary artery bypass grafting or percutaneous, transluminal coronary angioplasty); unstable angina; cerebrovascular accident, stroke, or transient ischemic attack; pacemaker; AF, flutter, or nonsustained or sustained ventricular tachycardia; orthostatic hypotension or orthostatic dizziness or lightheadedness, pulmonary arterial hypertension; sick sinus syndrome, second- or third-degree atrioventricular block; uncontrolled hypertension; congestive heart failure; personal or family history of sudden death or long QT syndrome; unexplained syncope or syncope within the last 3 years regardless of etiology.
* Immunization with a Coronavirus Disease (COVID-19) vaccine in the 14 days prior to the first study drug administration.
* Scheduled immunization with a COVID-19 vaccine during the study that, in the opinion of an Investigator, could potentially interfere with participant participation, participant safety, study results, or any other reason.
* Use of immunosuppressant in the 28 days or 5 half-lives (whichever is longer) prior to the first study drug administration.
* Major surgery with prolonged immobilization in the 28 days prior to the first study drug administration.
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
* Any clinically significant illness in the 28 days prior to the first study drug administration.
* Use of any over-the-counter or nutritional supplements in the last 7 days prior to the first study drug administration and during the study, that in the opinion of an Investigator would put into question the status of the participant as healthy.
* Use of any prescription drugs (including hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy.
* Use of St. John's Wort in the 28 days prior to the first study drug administration.
* Any history of tuberculosis.
* Hemoglobin value below the lower limit of the reference laboratory at Screening, unless deemed non-significant by the Investigator.
* Abnormal screening values in potassium, magnesium, alanine transaminase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase, alkaline phosphatase, total bilirubin, and direct bilirubin values, unless deemed non-significant by the Investigator
* Positive test result for urine alcohol and/or drugs of abuse at Screening or prior to the first drug administration.
* Current or history of alcohol or substance abuse, with the exception of being fully recovered with no use of alcohol or substances of abuse within the 12 months prior to Screening
* Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus antibody tests.
* Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
* History of prior administration of THRV-1268 or inclusion in a previous cohort for this clinical study.
* Treatment with any investigational product within 30 days or five half-lives of the drug (whichever is longer) prior to Screening.
* Unable or unwilling to adhere to the lifestyle and dietary requirements described in Section 5.5.
* Special diet or substantial changes in eating habits 1 month prior to Screening.
* Donation of 500 mL or more of blood (blood services, clinical studies, etc.) in the 56 days prior to Screening or donation of plasma within 7 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Evalute the safety and tolerability of a single oral dose | 7 days
  -Occurance of treatment emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetic THRV-1268 Tmax | From 0 to 24 hours
  Time to maximum observed plasma drug concentration
Pharmacokinetic THRV-1268 t1/2 | From 0 to 24 hours
  half-life
Pharmacokinetic THRV-1268 Cmax | From 0 to 24 hours
  Maximum observed plasma drug concentration
Pharmacokinetic THRV-1268 AUC0-t | From 0 to 24 hours
  Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable concentration
Evaluate and compare the bioavailability | From 0 to 24 hours
  To evaluate the relative bioavailability (Area under the plasma concentration versus time curve (AUC)) of THRV-1268 tablet relative to THRV-1268 API powder for oral

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided